CLINICAL TRIAL: NCT01785186
Title: A Multiple Arm, Multiple Stage, Phase 2, OL, Randomized, Controlled Trial to Evaluate 4 Treatment Regimens of SQ109, Increased Doses of Rifampicin, and Moxifloxacin in Adults With Newly Diagnosed, Smear-positive Pulmonary Tuberculosis
Brief Title: Evaluation of SQ109, High-dose Rifampicin, and Moxifloxacin in Adults With Smear-positive Pulmonary TB in a MAMS Design
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Hoelscher (Other)
Collaborators: Sequella, Inc. (Industry); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); German Federal Ministry of Education and Research (Other Government); Medical Research Council (Other Government); Radboud University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Michael Hoelscher, Prof., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PanACEA-MAMS-TB-01
Record Dates: First submitted 2012-12-17; First posted 2013-02-07 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-08

CONDITIONS: Tuberculosis, Pulmonary
Keywords: TB; Tuberculosis; MAMS - Multiple-arm, multiple-stage; Pulmonary; SQ109; High dose rifampicin; moxifloxacin
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis | interventions — Rifampin; Moxifloxacin; Isoniazid; Pyrazinamide; Ethambutol; Pyridoxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Arm 1 (R35) (Experimental): Arm 1 (R35): HR35ZE isoniazid, rifampicin 35 mg/kg, pyrazinamide, ethambutol
  Interventions: Drug: Rifampicin; Drug: isoniazid; Drug: pyrazinamide; Drug: ethambutol; Dietary Supplement: pyridoxine
- HRZQ (Experimental): Arm 2 (Q): HRZQ isoniazid, rifampicin standard, pyrazinamide, SQ109 300 mg
  Interventions: Drug: SQ109; Drug: Rifampicin; Drug: isoniazid; Drug: pyrazinamide; Dietary Supplement: pyridoxine
- HR20ZQ (Experimental): Arm 3 (R20Q): HR20ZQ isoniazid, rifampicin 20 mg/kg, pyrazinamide, SQ109 300 mg
  Interventions: Drug: SQ109; Drug: Rifampicin; Drug: isoniazid; Drug: pyrazinamide; Dietary Supplement: pyridoxine
- HR20ZM (Experimental): Arm 4 (R20M): HR20ZM isoniazid, rifampicin 20 mg/kg, pyrazinamide, moxifloxacin 400 mg
  Interventions: Drug: Rifampicin; Drug: isoniazid; Drug: pyrazinamide; Dietary Supplement: pyridoxine
- HRZE (Active Comparator): HRZE: Isoniazid, rifampicin standard, pyrazinamide, ethambutol
  Interventions: Drug: Rifampicin; Drug: Moxifloxacin; Drug: isoniazid; Drug: pyrazinamide; Drug: ethambutol; Dietary Supplement: pyridoxine

INTERVENTIONS:
Drug: SQ109 — SQ109 300 mg
  Arms: HR20ZQ; HRZQ
Drug: Rifampicin — Rifampicin 10 to 35 mg/kg
Drug: Moxifloxacin — Moxifloxacin 400mg
  Arms: HRZE
Drug: isoniazid — isoniazid 75 mg
Drug: pyrazinamide — pyrazinamide 400 mg
Drug: ethambutol — ethambutol 275 mg
  Arms: Arm 1 (R35); HRZE
Dietary Supplement: pyridoxine — pyridoxine 25 mg

SUMMARY:
This study is a multiple-arm, multiple-stage (MAMS), phase 2, open label, randomized, controlled clinical trial that will compare the efficacy and safety of four experimental four drug regimens with a standard control regimen in patients with smear positive, pulmonary tuberculosis (TB). Patients will be randomly allocated to the control or one of the four experimental regimens in the ratio 2:1:1:1:1. Experimental regimens will be given for 12 weeks. Thereafter, participants in the experimental arms will receive continuation phase treatment for 14 weeks containing standard-dose rifampicin and isoniazid. All participants will receive 25 mg of vitamin B6 (pyridoxine) with every dose of INH to prevent INH-related neuropathy. Interim analyses will be conducted during the trial for efficacy, with the aim of identifying experimental arms that perform below a pre-specified efficacy threshold; these arms will then be stopped from further recruitment.

Following the first scheduled interim analysis on March 3rd, the Trial Steering Committee (TSC) followed a recommendation of the independent data monitoring committee (IDMC) and has stopped the enrolment into two of the arms in the MAMS-TB trial: HRZQ and HR20ZQ, based on these arms not meeting the pre-specified gain in efficacy over control. Importantly, there was no safety concern that prompted stopping recruitment to these arms. They recommended that recruitment to arm 2 (HRZQ) and 3 (HR20ZQ) be terminated as there was insufficient evidence that these regimens could shorten treatment. Importantly, there was no evidence that either arm was inferior to standard treatment (the control arm) with regards to efficacy. There was, however, sufficient evidence that the other intervention arms HR35ZE and HR20ZM could shorten treatment to continue enrolling patients.

DETAILED DESCRIPTION:
This Phase II, multi-arm, multi-stage, open label, prospectively randomized, controlled clinical trial will compare the efficacy and safety of four experimental regimens with the control, standard treatment regimen in patients with smear positive, pulmonary tuberculosis (TB). There will be four experimental regimens. Participants will be randomly allocated to control or one of the four experimental intensive phase regimens in the ratio 2:1:1:1:1. The control and 4 experimental regimens are:

Control: HRZE isoniazid, rifampicin standard, pyrazinamide, ethambutol Arm 1: HRZQlow isoniazid, rifampicin standard, pyrazinamide, SQ109 150 mg Arm 2: HRZQhigh isoniazid, rifampicin standard, pyrazinamide, SQ109 300 mg Arm 3: HR20ZQhigh isoniazid, rifampicin 20 mg/kg, pyrazinamide, SQ109 300 mg Arm 4: HR20ZM isoniazid, rifampicin 20 mg/kg, pyrazinamide, moxifloxacin 400mg

Up to 372 participants will be randomized into this study, with 124 participants being randomized to the control arm and 62 participants to each experimental arm. With an expected loss to follow-up of 5%, the final power of the study to detect a hazard ratio of 1.8 for culture conversion to negative will be 90%, at the 5% significance level.

Participants will be randomised using a probabilistic minimisation algorithm based on site, baseline bacterial load as measured by GeneXpert MTB/RIF®, and HIV status. The allocated intensive phase of the four experimental arms will be administered daily for twelve weeks. During this time, participants will visit the study clinic on a weekly basis for sputum collection, safety monitoring and receipt of study medication. After the completion of the experimental treatment, participants in the experimental arms will receive daily standard continuation phase treatment for 14 weeks containing standard-dose RIF and INH to complete their TB treatment course. Participants in the control arm will receive eight weeks of intensive four-drug treatment (HRZE, followed by 18 weeks of the HR continuation phase treatment in line with the current WHO recommendations.

All participants will receive 25mg of Vitamin B6 (pyridoxine) with every dose of treatment in order to prevent INH-related neuropathy.

Interim analyses will be conducted during the trial for efficacy at predetermined times, with the aim of identifying experimental arms that perform below a pre-specified efficacy threshold. There will be no further recruitment to these arms.

ELIGIBILITY:
Inclusion Criteria

1. The patient has given free, signed written or witnessed oral informed consent for study participation prior to all trial-related procedures, including HIV testing if HIV serostatus is not known or the last documented negative is more than four weeks ago.
2. The patient has a diagnosis of pulmonary tuberculosis from a health clinic established by sputum smear and/or GeneXpert MTB/RIF® and/or chest X-ray.
3. An adequate sputum bacterial load is confirmed by a Ziehl-Neelsen stained smear in the study laboratory, done from concentrated sputum found at least 1+ on the IUATLD/WHO scale.
4. The patient has a valid rapid test result (GeneXpert MTB/RIF®) from the sputum positive for MTB complex, and indicating susceptibility to Rifampicin. This test must be done in the study laboratory.
5. The patient is aged at least 18 years at the day of informed consent.
6. The patient has a body weight in light clothing and without shoes of at least 35 kg, but not more than 90 kg.
7. Female patients of childbearing potential must have a negative serum pregnancy test, and consent to practise an effective method of birth control until week 26. Effective birth control for female patients has to include two methods, including methods that the patient's sexual partner(s) use. At least one must be a barrier method. Female patients are considered not to be of childbearing potential if they are post-menopausal with no menses for the last 12 months, or surgically sterile (this condition is fulfilled by bilateral oophorectomy, hysterectomy, and by tubal ligation which is done at least 12 months prior to enrolment).
8. Male patients must consent to use an effective contraceptive method, if their sexual partner(s) is/are of childbearing potential, and if they are not surgically sterile (see 6.). Contraception by male participants must be practised until at least week 24 to cover the period of spermatogenesis. Contraceptive methods used by male participants may include hormonal methods used by the partner(s).
9. The patient has a firm home address that is readily accessible for visiting and willingness to inform the study team of any change of address during trial participation, or will be compliant to study schedule, in the discretion of the investigator.

Exclusion Criteria

1. Circumstances that raise doubt about free, uncoerced consent to study participation (e.g. in a prisoner or mentally handicapped person)
2. Poor General Condition where delay in treatment cannot be tolerated or death within three months is likely.
3. The patient is pregnant or breast-feeding.
4. The patient has an HIV infection and is receiving antiretroviral treatment (ART), and/or is likely to require ART during the twelve weeks of experimental study treatment as per local guidelines.
5. The patient has a known intolerance to any of the study drugs, or concomitant disorders or conditions for which SQ109, rifampicin, moxifloxacin, or standard TB treatment are contraindicated.
6. The patient has an history or evidence of clinically relevant metabolic, gastrointestinal, neurological, psychiatric or endocrine diseases, malignancy, or any other condition that will influence treatment response, study adherence or survival in the judgement of the investigator, especially:

   clinically significant evidence of severe TB (e.g. miliary TB, TB meningitis. Limited lymph node involvement will not lead to exclusion); serious lung conditions other than TB or severe respiratory impairment in the discretion of the investigator; neuropathy, epilepsy or significant psychiatric disorder; uncontrolled and/or insulin-dependent diabetes; cardiovascular disease such as myocardial infarction, heart failure, coronary heart disease, uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure of ≥100 mmHg on two occasions), arrhythmia, or tachyarrhythmia; long QT syndrome (see criterion 9.), or family history of long QT syndrome or sudden death of unknown or cardiac-related cause; Plasmodium spp. parasitemia as indicated by thick blood smear or a positive rapid test present at screening; Alcohol or other drug abuse that is sufficient to significantly compromise the safety or cooperation of the patient, includes substances prohibited by the protocol, or has led to significant organ damage at the discretion of the investigator.
7. History of previous TB within the last five years.
8. Laboratory: at screening one or more of the following abnormalities were observed for the patient in screening laboratory: Serum amino aspartate transferase (AST) and/or serum alanine aminotransferase (ALT) activity >3x the upper limit of normal; Serum total bilirubin level >2.5 times the upper limit of normal; Creatinine clearance (CrCl) level lower than 30 mls/min; Complete blood count with hemoglobin level <7.0 g/dL; Platelet count <50,000/mm3; Serum potassium below the lower level of normal;
9. ECG findings in the screening ECG: QTcB and/or QTcF of >0.450 s; atrioventricular (AV) block with PR interval > 0.20 s; prolongation of the QRS complex over 120 milliseconds; other changes in the ECG that are clinically relevant as per discretion of the investigator.
10. The patient has had treatment with any other investigational drug within 1 month prior to enrolment, or enrolment into other clinical (intervention) trials is planned during week 1-26
11. Previous anti-TB treatment: the patient has had previous treatment with drugs active against M. tuberculosis within the last 3 months, including but not limited to INH, EMB, RIF, PZA, amikacin, cycloserine, rifabutin, streptomycin, kanamycin, para-aminosalicylic acid, rifapentine, thioacetazone, capreomycin, fluoroquinolones, thioamides.
12. QT prolonging medications: Administration within 30 days prior to study start, anticipated administration during the study period, or during the 12 weeks of experimental treatment, of any QT-prolonging agents such as, but not limited to, azithromycin, bepridil chloroquine, chlorpromazine, cisapride, cisapride, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, lumefantrine, mefloquine, mesoridazine, methadone, moxifloxacin, pentamidine, pimozide, procainamide, quinidine, quinine, roxithromycin, sotalol, sparfloxacin, terfenadine, thioridazine. Exceptions may be made for participants who have received 3 days or less of one of these drugs or substances, if there has been a wash-out period equivalent to at least 5 half-lives of that drug or substance.

    Patients who have ever received amiodarone will be excluded from study participation.
13. CYP 450 inducers/inhibitors: administration within 30 days prior to dosing, or planned administration until the end of week 12, of any drug(s) or substance(s) known to be strong inhibitors or inducers of cytochrome P450 enzymes, or specific inhibitors/inducers of SQ109-metabolizing enzymes as Exceptions may be made for subjects that have received 3 days or less of one of these drugs or substances, if a wash-out period equivalent to at least 5 half-lives of that drug or substance prior to study treatment is granted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hoelscher, MD, Study Chair — Klinikum of the University of Munich; Martin Boeree, MD, Principal Investigator — Radboud University Medical Center
Locations (7):
- South Africa (4):
  - TASK Applied Science, Bellville
  - University of Cape Town, Centre for Tuberculosis Research Innovation, Cape Town
  - Wits Health Consortium, Johannesburg
  - The Aurum Institute for Health Research, Johannesburg
- Tanzania (3):
  - Ifakara Health Institute, Bagamoyo
  - NIMR - Mbeya Medical Research Programme, Mbeya
  - Kilimanjaro Christian Medical Centre (KCMC) / Kilimanjaro Clinical Research Institute (KCRI) (with affiliated field sites such as Kibong'oto National Tuberculosis Hospital Same, Mererani, Chekereni and Mawenzi Regional Hospital), Moshi

REFERENCES:
- [Derived] Zhang N, Savic RM, Boeree MJ, Peloquin CA, Weiner M, Heinrich N, Bliven-Sizemore E, Phillips PPJ, Hoelscher M, Whitworth W, Morlock G, Posey J, Stout JE, Mac Kenzie W, Aarnoutse R, Dooley KE; Tuberculosis Trials Consortium (TBTC) and Pan African Consortium for the Evaluation of Antituberculosis Antibiotics (PanACEA) Networks. Optimising pyrazinamide for the treatment of tuberculosis. Eur Respir J. 2021 Jul 20;58(1):2002013. doi: 10.1183/13993003.02013-2020. Print 2021 Jul. PMID 33542052
- [Derived] Boeree MJ, Heinrich N, Aarnoutse R, Diacon AH, Dawson R, Rehal S, Kibiki GS, Churchyard G, Sanne I, Ntinginya NE, Minja LT, Hunt RD, Charalambous S, Hanekom M, Semvua HH, Mpagama SG, Manyama C, Mtafya B, Reither K, Wallis RS, Venter A, Narunsky K, Mekota A, Henne S, Colbers A, van Balen GP, Gillespie SH, Phillips PPJ, Hoelscher M; PanACEA consortium. High-dose rifampicin, moxifloxacin, and SQ109 for treating tuberculosis: a multi-arm, multi-stage randomised controlled trial. Lancet Infect Dis. 2017 Jan;17(1):39-49. doi: 10.1016/S1473-3099(16)30274-2. Epub 2016 Oct 26. PMID 28100438

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HRZQ | Arm 1 (R35) | HR20ZQ | HR20ZM | HRZE
Started | 59 | 63 | 57 | 63 | 123
Completed | 53 | 57 | 52 | 58 | 117
Not Completed | 6 | 6 | 5 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HRZQ | Arm 1 (R35) | HR20ZQ | HR20ZM | HRZE | Total
Number analyzed (Participants) | 59 | 63 | 57 | 63 | 123 | 365
Age, Customized [Median (Inter-Quartile Range); unit: years] | 32 [25 to 40] | 33 [23 to 40] | 34 [27 to 41] | 31 [24 to 38] | 34 [26 to 41] | 32.9 [23.8 to 40.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 12 | 24 | 29 | 107
  Male | 38 | 42 | 45 | 39 | 94 | 258
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 50 | 51 | 50 | 48 | 101 | 300
  White | 0 | 1 | 1 | 0 | 0 | 2
  More than one race | 9 | 11 | 6 | 15 | 19 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 3
HIV Positive Participants [Number; unit: participants] | 5 | 4 | 3 | 3 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Sputum Culture Conversion (2 Negative Cultures) Using Liquid Media
Description: From enrollment, the time to stable culture conversion (2 consecutive negative weekly cultures) in liquid media.
Time Frame: 0 - 12 weeks
Population: Modified intention to treat analysis
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Arm 1 (R35) | HRZQ | HR20ZQ | HR20ZM | HRZE
Number analyzed (Participants) | 63 | 58 | 56 | 63 | 123
days | 48 [34 to 69] | 63 [48 to 83] | 66 [41 to 83] | 55 [41 to 69] | 62 [41 to 83]

2. Secondary Outcome: Frequency of Adverse Events
Description: All Adverse Events (AE), and AEs considered to be drug-related will coded using standard AE dictionaries.
Time Frame: 0 - 12 weeks
Measure: Number; unit: participants
Arm/Group | Arm 1 (R35) | HRZQ | HR20ZQ | HR20ZM | HRZE
Number analyzed (Participants) | 63 | 58 | 56 | 63 | 123
participants
  Number of Patients with at least 1 AE | 53 | 49 | 42 | 49 | 92
  Number of patients with at least 1 SAE | 4 | 4 | 5 | 4 | 6

3. Secondary Outcome: Mycobacteriology Identification and Characterization by PCR and MIC
Description: Cultures grown from the screening period, and the last sputum sample with mycobacteriological growth will be assessed as follows:
  * Identification of M. tuberculosis complex and RIF resistance by PCR (GeneXpert MTB/RIF®),
  * First-line drug susceptibility testing of the M. tuberculosis isolates using the MGIT system for sensitivity to rifampicin; isoniazid, pyrazinamide, moxifloxacin or ethambutol.
  * Minimum inhibitory concentrations (MIC) of SQ109, rifampicin and moxifloxacin.
  * Typing of the infecting strain(s) by molecular methods.
Time Frame: 0 - 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Pharmacokinetics Including AUC, Cl, t1/2, Vd, and Protein Binding
Description: Pharmacokinetic parameters will be assessed for rifampicin, moxifloxacin and SQ109:
  * area under the plasma concentration curve from dosing to the end of the dosing interval (AUC 0-24) (in h*ng/mL)
  * the observed maximum concentration (Cmax( (in ng/mL)
  * time to reach Cmax (Tmax)(in hours)
  * the minimum observed plasma concentration 24 hours following the last dose (Cmin) (in hours),
  * clearance (Cl) (in mL/minute),
  * volume of distribution (Vd) (in L),
  * elimination half-life (T1/2,) (in hours)
  * free (protein-unbound) fraction (for rifampicin only) (in percent).
Time Frame: 0 - 12 weeks
Population: Pharmacokinetic population
Measure: Geometric Mean (Full Range); unit: Rifampicin AUC(mg*h/l)
Arm/Group | HRZQ | Arm 1 (R35) | HR20ZQ | HR20ZM | HRZE
Number analyzed (Participants) | 19 | 20 | 19 | 19 | 19
Rifampicin AUC(mg*h/l) | 17.4 [4.3 to 45.3] | 170 [103 to 266] | 68.3 [38.5 to 149] | 57.8 [15 to 121] | 24.2 [11.9 to 52.5]

5. Secondary Outcome: Pharmacodynamics Including AUC0-24/MIC (h*ng/mL) and Cmax/MIC (ng/mL)
Description: By combining pharmacokinetic parameters and MIC values (see below), the pharmacodynamic indices AUC0-24/MIC (h*ng/mL) and Cmax/MIC (ng/mL) will be calculated for individual patients for experimental drugs administered. Pharmacokinetic parameters and pharmacodynamic indices will be related to efficacy and safety/tolerability endpoints.
Time Frame: 0 - 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Time to First Negative Culture on Liquid and Solid Media
Description: Time to a convert to a single negative culture on liquid and solid media
Time Frame: 0 - 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Proportion of Negative Sputum Cultures
Description: Proportion of patients converting to negative sputum culture (2 consecutive weekly cultures) in liquid and solid media
Time Frame: 0 - 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Rate of Change in Time to Positivity
Description: Rate of change in time to positivity in BD MGIT 960® liquid culture
Time Frame: 0 - 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Rate of Change in Quantitative PCR During Therapy
Description: GeneXpert MTB/RIF (Xpert) quantitative PCR results (counts per week
Time Frame: 0 - 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Occurence of Treatment Failure (Relapse or Emergence of Drug-resistance)
Description: Frequency of treatment failures (number of patients with relapse and/or development of drug resistance) will be recorded
Time Frame: 0 - 12 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Changes in Baseline Laboratory Safety Parameters During Treatment and Follow-up
Description: Frequency tables will be generated for visual acuity tests, 12 lead ECGs, clinical chemistry metrics, haematology, and urinalysis
Time Frame: 0 - 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | HRZQ | Arm 1 (R35) | HR20ZQ | HR20ZM | HRZE
Serious Adverse Events (participants affected / at risk) | 4/59 | 4/63 | 5/57 | 4/63 | 6/123
Other Adverse Events (participants affected / at risk) | 49/59 | 53/63 | 42/57 | 49/63 | 92/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HRZQ (N=59) | Arm 1 (R35) (N=63) | HR20ZQ (N=57) | HR20ZM (N=63) | HRZE (N=123)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychosis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis of ankles (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
left pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intrahepatic cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parasuicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Resiratory insufficiency secondary to psnumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
haemoptysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral fractures due to post motor vehicle accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Community accuired pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multi drug resistant TB (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fever - hospitalization (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hyper osmolar hyperglycaemia state (diabetic melitus) grade 4 (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parasuicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HRZQ (N=59) | Arm 1 (R35) (N=63) | HR20ZQ (N=57) | HR20ZM (N=63) | HRZE (N=123)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abcess of eyelid (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 6 (6)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 1 (2) | 2 (2) | 2 (2)
Alcoholic liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (8) | 8 (8) | 6 (7) | 10 (10) | 18 (19)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 3 (3)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood albumine decreased (Investigations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Body tinea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (5) | 4 (4) | 2 (2) | 6 (6)
Conjunctival discolouration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis allergic (Immune system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 6 (7)
Dental caries (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 2 (2) | 2 (2) | 5 (5) | 4 (4)
Drug eruption (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
drug induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
duodenitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0)
Eye irrritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
fungal skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GGT increased (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
gastroentertitis bacterial (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
goitre (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
haemoptysis (Blood and lymphatic system disorders) | 7 (10) | 3 (3) | 4 (4) | 5 (5) | 7 (10)
haemarrhoids (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
headache (General disorders) | 6 (8) | 5 (5) | 4 (4) | 4 (6) | 11 (11)
heart rate increased (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hepatic enzyme increased (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
herpes simplex (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
herplex zoster (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
hypercholsterolaemia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hyperglycaemia (Endocrine disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 4 (4)
Influenza (Infections and infestations) | 5 (5) | 4 (4) | 1 (1) | 4 (4) | 7 (7)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 2 (2) | 4 (4) | 4 (5) | 2 (2) | 2 (2)
Liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Malaria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 4 (4) | 2 (2) | 2 (2)
Myopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 7 (7) | 9 (9) | 8 (8) | 7 (9) | 7 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Night sweats (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic neuritis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Pain in face (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericarditis tuberculous (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post thrombotic syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-tussive vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pregnancy test false positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 11 (14) | 5 (6) | 9 (9) | 17 (18)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 3 (3) | 3 (3) | 2 (3) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 6 (6) | 5 (5) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 | 3 (4)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 2 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis seasonal (Immune system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Serum ferritin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Tenderness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tinea capitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 2 (2) | 4 (6)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urogenital infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Visual acuity reduced transiently (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (6) | 11 (11) | 8 (8) | 8 (9) | 15 (16)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 2 (3)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other